CLINICAL TRIAL: NCT06046482
Title: Phase II Trial of Magrolimab and Cetuximab With Pembrolizumab or Docetaxel for Recurrent/Metastatic Head Neck Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0903; NCI-2023-07199 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Head Neck; Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; magrolimab; Cetuximab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Participants will receive magrolimab and cetuximab along with pembrolizumab.
  Interventions: Drug: Pembrolizumab; Drug: Magrolimab; Drug: cetuximab
- Cohort B (Experimental): Participants will receive magrolimab and cetuximab along with docetaxel.
  Interventions: Drug: Magrolimab; Drug: cetuximab; Drug: Docetaxel

INTERVENTIONS:
Drug: Pembrolizumab — Given by IV (vein)
  Other Names: KEYTRUDA®
  Arms: Cohort A
Drug: Magrolimab — Given by IV (vein)
Drug: cetuximab — Given by IV (vein)
  Other Names: ERBITUX
Drug: Docetaxel — Given by IV (vein)
  Arms: Cohort B

SUMMARY:
To learn if magrolimab, along with a combination of commercially-available drugs (cetuximab, pembrolizumab, and docetaxel) can help to control HNSCC in combination with other drugs. The safety of magrolimab will also be studied.

DETAILED DESCRIPTION:
Primary Objectives:

-Objective response rate (ORR) per RECIST v1.1

Secondary Objectives:

* Adverse events rates per CTCAE V5.0 (appendix)
* Duration of response (DOR)
* Progression free survival (PFS) per RECIST v1.1
* Overall survival (OS) per RECIST v1.1

Exploratory Objectives:

-Assessment of blood and tissue-based biomarkers predictive of response to therapy

ELIGIBILITY:
Inclusion Criteria:

All patients must meet all of the following inclusion criteria to be eligible for participation in this study:

1. Patient must have a diagnosis of recurrent or metastatic oropharynx, oral cavity, hypopharynx, or larynx squamous cell carcinoma (HNSCC), not amenable to curative-intent local therapy with known PD-L1 CPS determined by an FDA-approved test. Patients with unknown primary squamous cell carcinoma presumed from the head and neck are also eligible upon discussion with study principal investigator.
2. Patient has provided informed consent.
3. Patient is willing and able to comply with clinic visits and procedures outlined in the study protocol.
4. Male or female ≥ 18 years of age
5. ECOG performance status of 0 or 1
6. Laboratory measurements, blood counts:

   1. Hemoglobin ≥ 9 g/dL within 24 hours prior to initial dose of study treatment. Red blood cell transfusions are permitted to meet the hemoglobin inclusion criteria, within limits set per exclusion criterion 6.
   2. Absolute neutrophil count ≥ 1.2 x 109/mL
   3. Platelets ≥ 100 x 109/mL
7. Laboratory measurements, renal function:

   Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or if elevated, a calculated glomerular filtration rate > 40 mL/min/1.73m2 per CKD-EPI equation.
8. Laboratory measurements, hepatic function:

   1. AST and ALT ≤ 2.5 x ULN or ≤ 5 x ULN in patients with liver metastases
   2. Total bilirubin ≤ 1.5 x ULN or ≤ 3.0 x ULN and primarily unconjugated if patient has a documented history of Gilbert's syndrome or genetic equivalent
9. Laboratory measurements, coagulation function:

   1. International normalized ratio or prothrombin time (PT) ≤ 1.5 x ULN unless patient is receiving anticoagulation therapy, as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use for anticoagulants
   2. Activated partial thromboplastin time or PTT ≤ 1.5 x ULN unless patient is receiving anticoagulation therapy, as long as PT or PTT is within therapeutic range of intended use for anticoagulants
10. Female patients with reproductive potential must practice two effective contraceptive measures for the duration of study drug therapy and for at least 6 months after completion of study therapy. The two birth control methods can be either two barrier methods or a barrier method plus a hormonal method to prevent pregnancy. The following are considered adequate barrier methods of contraception: diaphragm, condom, copper intrauterine device, sponge, or spermicide. Appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents).
11. Male patients who are sexually active with women with reproductive potential must agree to use contraception for the duration of treatment and for at least 6 months after completion of study therapy.
12. Measurable disease according to RECIST, version 1.1
13. Patients must be willing to provide baseline tumor tissue from a core or excisional biopsy (fine needle aspirate is not adequate). A newly obtained biopsy (within 90 days prior to study treatment start) is strongly preferred, but an archival sample is acceptable.
14. Absence of active auto-immune disease or any other contra-indication to pembrolizumab, cetuximab, docetaxel or magrolimab

    Cohort A:

    In addition to meeting the inclusion criteria for all patients, patients who are enrolled into Cohort A must fulfill the following cohort-specific inclusion criteria:
15. PD-L1 CPS must be ≥ 1
16. Patients should not have had prior systemic therapy administered in the recurrent or metastatic setting. Systemic therapy that was completed more than 3 months prior to signing consent if given as part of multimodal treatment for locally advanced disease is allowed.
17. Patients could have received anti-PD1 or anti-PD-L1 in the neoadjuvant or adjuvant setting as part of a clinical trial, as long as the patient has not progressed during it and there has been at least a 6 months disease-free interval since last administration of anti-PD1 or anti-PD-L1 in the curative intent setting.

Cohort B:

In addition to meeting the inclusion criteria for all patients, patients who are enrolled into Cohort B must fulfill the following cohort-specific inclusion criterion:

17) Patients must have received at least 1 and no more than 2 lines of prior systemic anticancer therapy in the recurrent/metastatic setting not including docetaxel but including anti-PD1. Patients must have progressed on anti-PD1 (radiographically or clinically) or developed intolerable adverse events attributed to anti-PD1 that lead to treatment discontinuation and eventual disease progression. Patients with contra-indications to anti-PD1 are also eligible.

Exclusion Criteria:

Patients who meet any of the following exclusion criteria are not eligible to be enrolled in this study:

1. Prior radiation therapy (or other nonsystemic therapy) within 2 weeks prior to enrollment
2. Patient has not fully recovered (ie, ≤ Grade 1 at baseline) from AEs due to a previously administered treatment.

   1. Note: Patients with ≤ Grade 2 neuropathy, alopecia, or laboratory values in inclusion criteria 5 through 8 are exceptions to this criterion and may qualify for the study.
   2. Note: If a patient received major surgery, he or she must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
3. Active CNS disease (patients with asymptomatic and stable, treated CNS lesions who have been off corticosteroids, radiation, or other CNS-directed therapy for at least 4 weeks are not considered active)
4. Red blood cell transfusion dependence, defined as requiring more than 2 units of packed RBC transfusions during the 4-week period prior to screening. Red blood cell transfusions are permitted during the screening period and prior to enrollment to meet the hemoglobin inclusion criterion.
5. History of hemolytic anemia, autoimmune thrombocytopenia, or Evans syndrome in the last 3 months
6. Known inherited or acquired bleeding disorders
7. Prior treatment with CD47 or SIRPα-targeting agents
8. Prior anticancer therapy including, but not limited to, chemotherapy, immunotherapy, or investigational agents within 4 weeks prior to magrolimab treatment
9. Life expectancy of less than 3 months and/or rapidly progressing disease (eg, tumor bleeding, uncontrolled tumor pain) in the opinion of the treating investigator
10. Diagnosis of immunodeficiency or receipt of systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study therapy. Corticosteroid use as a premedication for biopsy, allergic reactions or for prophylactic management of AEs related to the chemotherapies specified in the protocol is allowed. The use of physiologic doses of corticosteroids may be approved with approval by the sponsor.
11. Active autoimmune disease that has required systemic treatment in the past 2 years (ie, use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
12. Prior allogeneic tissue/solid organ transplant
13. Current participation in another interventional clinical study
14. History of previous malignancy other than malignancy treated with curative intent and with no evidence of active disease ≥ 2 years before the first dose of the study drugs and of low potential risk for recurrence. Patients with the following diagnoses represents an exception and may enroll:

    1. Non-melanoma skin cancers with no current evidence of disease
    2. Melanoma in situ with no current evidence of disease
    3. Localized cancer of the prostate with prostate-specific antigen of <1 ng/mL
    4. Treated or localized well-differentiated thyroid cancer
    5. Treated cervical carcinoma in situ
    6. Treated ductal/lobular carcinoma in situ of the breast
15. Evidence of uncontrolled, active infection, requiring systemic anti-bacterial, anti-viral or anti-fungal therapy ≤ 10 days prior to administration of investigational product. Patients with known hepatitis B, hepatitis C (HCV), or HIV infection could go on study provided the viral load is undetectable at Screening.
16. Significant disease or medical conditions, as assessed by the investigator and sponsor, that would substantially increase the risk-benefit ratio of participating in the study. This includes, but is not limited to, acute myocardial infarction within the last 6 months, unstable angina, uncontrolled diabetes mellitus, significant active infections, and congestive heart failure New York Heart Association Class III-IV
17. Female subjects who are pregnant or breast-feeding
18. Known hypersensitivity to any of the study drugs, the metabolites, or formulation excipient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renata Ferrarotto, M D, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Anti-PD1 naïve, treatment with Magrolimab, Cetuximab, and Pembrolizumab and Cohort A Maintenance
  Anti-PD1 naïve, magro IV QW/cetux IV QW/pembro IV Q3W
- Cohort B: Anti-PD1 refractory, treatment with Magrolimab, Cetuximab and Docetaxel
  Anti-PD1 refractory magro IV QW/cetux IV QW/docetaxel IV QW
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 1 | 3
Completed | 1 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) per RECIST v1.1. Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v.1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >= 30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient growth to qualify for PD; Progressive Disease (PD), >= 20% increase in the sum of the longest diameter with an absolute increase of at least 5 mm or the appearance of new lesions
Time Frame: 140 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 1 | 3
Participants
  Partial Response (PR) | 1 | 0
  Stable Disease (SD) | 0 | 3

2. Secondary Outcome: Number of Treatment-Emergent Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0
Description: Adverse events (AEs) are categorized as follows: Treatment-Emergent Adverse Events (TEAEs), which refer to any AEs that arise or worsen in severity after the initiation of treatment with the study product; and Treatment-Related Adverse Events (TRAEs), defined as TEAEs that are considered possibly, probably, or definitely related to the treatment. Adverse Events were graded 1 to 5 via CTAE 5.0 guidelines. All AEs, whether serious or non-serious, will be captured from the time of the first administration of the investigational agent until 30 days following the last dose of study drug or until the initiation of alternative anticancer therapy
Time Frame: 145 days
Measure: Number; unit: Treatment-Emergent Adverse Events TEAEs
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 1 | 3
Treatment-Emergent Adverse Events TEAEs
  Grade 3 : Definite | 0 | 1
  Grade 3 : Possible | 0 | 2
  Grade 3 : Probable | 0 | 0
  Grade 3 : Unlikely | 0 | 0
  Grade 3 : Unrelated | 1 | 0
  Grade 2 : Definite | 1 | 2
  Grade 2 : Possible | 3 | 2
  Grade 2 : Probable | 0 | 3
  Grade 2 : Unlikely | 0 | 0
  Grade 2 : Unrelated | 3 | 1
  Grade 1 : Definite | 1 | 8
  Grade 1 : Possible | 8 | 17
  Grade 1 : Probable | 2 | 5
  Grade 1 : Unlikely | 3 | 10
  Grade 1 : Unrelated | 9 | 5

3. Secondary Outcome: Duration of Response (DOR)
Description: Time (the duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented.
Time Frame: 2 weeks and 1 day
Population: Cohort A - participant withdrew consent after 15 days. Cohort B -- no patients in cohort B achieved a PR.
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With Progression Free Survival (PFS) and/or Death
Description: Progression free survival (PFS) per RECIST v1.1. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) as a 20% increase in the sum of the longest diamester of target lesions, a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 4 months and 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 1 | 3
Participants
  Disease progression | 0 | 1
  Death on study | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time the first patient signed consent until the last patient has completed the observation period as designated by the protocol (pg. 45: All Aes whether serious or non-serious, will be captured from the time of the first administration of the investigational agent until 30 days following the last dose of study drug or until the initiation of alternative anticancer therapy): 145 days
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/3
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=1) | Cohort B (N=3)
Colitis (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=1) | Cohort B (N=3)
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 1
Alkaline phosphatase increased (Investigations) | 1 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 3
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Creatinine Increased (Investigations) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eye Pain (Eye disorders) | 1 | 0
Fatigue (General disorders) | 0 | 2
Flushing (Vascular disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagenesemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2
Insomnia (General disorders) | 1 | 0
Investigations, other specify (Investigations) | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 0 | 2
Neutrophil count decreased (Investigations) | 1 | 1
Paresthesia (Nervous system disorders) | 0 | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 1
Platelet Count Decreased (Investigations) | 1 | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 | 3
Restlessness (General disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 1 | 1
Urine discoloration (Renal and urinary disorders) | 1 | 0
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT06046482/Prot_SAP_001.pdf
  • Informed Consent Form (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT06046482/ICF_000.pdf